CLINICAL TRIAL: NCT03123731
Title: iSTEP - an mHealth Physical Activity and Diet Intervention for Persons With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Brook Henry, Associate Project Scientist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 161347; 5R01AG074808 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: HIV/AIDS
Keywords: physical activity; diet; mHealth; Fitbit; neurocognition; text messaging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): Participants will wear a Fitbit but will not receive any additional elements of the iSTEP intervention.
  Interventions: Behavioral: Control Arm
- iSTEP PA intervention (Experimental): Participants will wear a Fitbit and receive interactive daily text messages that are designed to motivate moderate physical activity (PA) and reduce sedentary behavior, including setting weekly goals to increase average daily step counts.
  Interventions: Behavioral: iSTEP
- iSTEP PA and diet intervention (Experimental): Participants will wear a Fitbit and receive interactive daily text messages that are designed to motivate moderate physical activity (PA), reduce sedentary behavior, and promote adherence to a Mediterranean-style diet. Participants will also be administered diet counseling from a registered dietitian and receive weekly feedback on both physical activity and diet behaviors.
  Interventions: Behavioral: iSTEP

INTERVENTIONS:
Behavioral: Control Arm — Wearing Physical Activity Monitor
  Arms: Control Arm
Behavioral: iSTEP — Physical Activity Intervention
  Arms: iSTEP PA intervention
Behavioral: iSTEP — Physical Activity and Diet Intervention
  Arms: iSTEP PA and diet intervention

SUMMARY:
HIV is associated with a pattern of neurocognitive deficits, metabolic dysfunction, and an elevated risk for cardiovascular disease (CVD), phenomena that remain untreated despite the use of medications to control the disease. This proposal will examine the effect of a personalized, automated, interactive mobile phone text message intervention (iSTEP) designed to increase moderate physical activity (PA), decrease sedentary behavior (SB), and promote a healthy Mediterranean-style diet (MedDiet) in persons living with HIV (PLWH). The investigators propose that participants who receive the iSTEP intervention will increase the amount of physical activity, improve their diet, show a reduction in risk factors for CVD, and exhibit improved neurocognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* HIV infection documented at the University of California, San Diego (UCSD) HIV Neurobehavioral Research Program (HNRP) or assessed by an HIV test at screening
* proficient in English
* physically capable of participating in moderate PA as screened by the Physical Activity Readiness Questionnaire
* consent from primary care physician to participate in the study
* able to consume walnuts - no nut allergies

Exclusion Criteria:

* any physical conditions that would prevent moderate physical activity or where moderate physical activity would represent a health risk for the individual, including a history of myocardial infarction or stroke
* unwillingness or inability to participate in daily text messaging
* tree nut allergy that would prevent walnut consumption or other food restrictions that would prevent participation in the Mediterranean-style diet intervention (e.g., unable to eat fish or use olive oil for cooking).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brook L Henry, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- HIV Neurobehavioral Research Program, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henry BL, Quintana E, Moore DJ, Garcia J, Montoya JL. Focus groups inform a mobile health intervention to promote adherence to a Mediterranean diet and engagement in physical activity among people living with HIV. BMC Public Health. 2019 Jan 22;19(1):101. doi: 10.1186/s12889-018-6386-5. PMID 30669986

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Started | 32 | 35 | 33
Completed | 23 | 21 | 26
Not Completed | 9 | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention | Total
Number analyzed (Participants) | 32 | 35 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 51 (15) | 52 (13) | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 28 | 30 | 28 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 5 | 5 | 4 | 14
  White | 21 | 21 | 26 | 68
  More than one race | 1 | 4 | 0 | 5
  Unknown or Not Reported | 4 | 3 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 35 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity - Total Steps Recorded During 24 Weeks
Description: Total number of steps recorded by the Fitbit over 24 weeks. Zero is the minimum and there is no maximum. Higher scores (steps) indicates a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 25 | 24 | 27
steps | 1345700 (99288) | 1686395 (187679) | 1684843 (137606)

2. Secondary Outcome: Physical Activity - Change in Average Daily Steps Per Day Between Week 1 and Week 24
Description: This is the change in average daily steps comparing the beginning (Week 1) and end (Week 24) of the intervention. A higher number is a positive outcome, indicated an increase in steps during the study. A negative number is a worse outcome, indicating a decline in steps during the intervention. Zero is the minimum and there is no maximum.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: steps/day
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 23 | 19 | 25
steps/day | -1504 (620) | 1667 (1086) | -685 (921)

3. Secondary Outcome: Average Steps Per Day During the 24-week Intervention
Description: This measure reports the average daily steps per day during the entire intervention (over 24 weeks). A higher number of steps indicates greater physical activity and is a positive outcome. A lower number of daily steps indicates lower physical activity. Zero is the minimum and there is no maximum.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: steps/day
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 24 | 22 | 27
steps/day | 8081 (588) | 10850 (1179) | 10015 (787)

4. Secondary Outcome: C-reactive Protein
Description: The change in C-reactive protein between baseline and the follow-up visit after the 24-week intervention. Higher numbers indicate that inflammation increased over time, a worse outcome. Lower numbers indicate less inflammation, a better outcome.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 18 | 13 | 17
pg/ml | -289405 (682583) | -63545 (603429) | -239997 (729441)

5. Secondary Outcome: Change in Total Cholesterol.
Description: This measures the change in total plasma cholesterol between the baseline visit and the 24-week follow-up visit. A decrease in cholesterol is healthy, while an increase is unhealthy.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 21 | 18 | 21
mg/dL | 2.14 (4.56) | 17.83 (11.77) | 10.04 (4.72)

6. Secondary Outcome: Level of GPLD1 (Phosphatidylinositol-glycan-specific Phospholipase D) Enzyme at the Baseline Visit
Description: This measures the plasma level of GPLD1 at the baseline study visit before the 24-week intervention. Higher levels are hypothesized to be positive and associated with better health and lower inflammation.The minimum level is zero and there is no maximum limit.
Time Frame: 1 day baseline visit
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 19 | 12 | 20
pg/ml | 190278 (12179) | 196997 (17343) | 168417 (13811)

7. Secondary Outcome: Change in GPLD1 (Phosphatidylinositol-glycan-specific Phospholipase D) Enzyme Between the Baseline and 24-week Visit
Description: This measures the change in GPLD1 between the baseline and 24-week visit after the study intervention. An increase in GPLD1 is hypothesized to associate with health benefits, while a decrease is a negative outcome.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 19 | 11 | 20
pg/ml | 14497 (12720) | -36496 (21248) | 29674 (15927)

8. Secondary Outcome: Association Between Physical Activity (PA) and GPLD1 (Phosphatidylinositol-glycan-specific Phospholipase d) at Baseline
Description: This measures the correlation (Pearson r) between GPLD1 (measured on one 1 day) and participant PA (assessed by average daily steps for 1 week) at the baseline before the 24-week intervention. A positive number indicates that higher GPLD1 was associated with greater PA. A negative number indicates that higher GPLD1 associates with lower PA. The minimum value is -1. The maximum value is +1.
Time Frame: 1 week
Measure: Number; unit: Pearson's r
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 19 | 14 | 20
Pearson's r | -0.175 | -4.06 | -0.05

9. Secondary Outcome: Association Between the Change in Physical Activity (PA) and Change in GPLD1 (Phosphatidylinositol-glycan-specific Phospholipase d) Between the Baseline Visit and 24-week Visit After the Intervention
Description: This measures the correlation (Pearson r) between the change in GPLD1 across the baseline and 24-week visits and the change in PA (average daily steps) between the first week (Week 1) and last week (Week 24) of the study. A positive number indicates that an increase in GPLD1 associated with an increase in PA over time, a negative number indicates the opposite. The minimum value is -1. The maximum value is +1.
Time Frame: 24 weeks
Measure: Number; unit: Pearson's r
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 19 | 13 | 19
Pearson's r | -0.354 | 0.147 | 0.363

10. Secondary Outcome: Association Between Cognitive Performance (Executive Function) and GPLD1 (Phosphatidylinositol-glycan-specific Phospholipase d) at the 24-week Visit After the Intervention
Description: This measures the correlation (Pearson r) between GPLD1 and executive function (measured by T score) at the 24-week visit after the intervention. A positive number indicates that higher GPLD1 associates with better executive function. A negative number indicates that higher GPLD1 associates with worse cognition (lower T score). The minimum value is -1. The maximum value is +1.
Time Frame: 1 day at the end of the 24-week intervention
Measure: Number; unit: Pearson's r
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 20 | 14 | 19
Pearson's r | 0.332 | 0.226 | 0.213

11. Secondary Outcome: Association Between the Change in Inflammation (C-reactive Protein, or CRP) and Change in GPLD1 (Phosphatidylinositol-glycan-specific Phospholipase d) Between the Baseline and 24-week Visits.
Description: This measures the correlation (Pearson r) between the change in CRP and the change in GPLD1 across the baseline and 24-week visits. A positive number indicates that an increase in GPLD1 associated with an increase in CRP (higher inflammation). A negative number indicates that an increase in GPLD1 associated with a decrease in CRP (lower inflammation). The minimum value is -1. The maximum value is +1.
Time Frame: 24 weeks
Measure: Number; unit: Pearson's r
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
Number analyzed (Participants) | 18 | 13 | 17
Pearson's r | -0.401 | -0.422 | 0.174

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the 24-week (6-month) study intervention for each participant.
Arm/Group | Control Arm | iSTEP PA Intervention | iSTEP PA and Diet Intervention
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 9/32 | 10/35 | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=32) | iSTEP PA Intervention (N=35) | iSTEP PA and Diet Intervention (N=33)
Myocardial infarction (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=32) | iSTEP PA Intervention (N=35) | iSTEP PA and Diet Intervention (N=33)
minor muscle soreness (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03123731/Prot_SAP_000.pdf